CLINICAL TRIAL: NCT04392453
Title: Upper Limb Robotic Rehabilitation in Stroke Survivors Using a Portable Device During the COVID-19 Outbreak. A Feasibility Study
Brief Title: Upper Limb Robotic Rehabilitation During COVID-19 Outbreak
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Irene Giovanna Aprile, MD, PhD, Fondazione Don Carlo Gnocchi Onlus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDG_Icone
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Stroke
Keywords: rehabilitation; stroke; upper extremity; robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic therapy (Experimental): Upper limb robotic rehabilitation by means of the portable robot Icone.
  Interventions: Device: Robotic therapy

INTERVENTIONS:
Device: Robotic therapy — The treatment with the robot Icone will include 30 sessions, each session lasting 45 minutes, with a frequency from three to five times a week. The treatment will be provided in the patient's room. Patients will execute upper limb movement involving elbow flexion-extension, shoulder protraction-retraction, internal-external rotation, flexion-extension, and abduction-adduction. Visual and auditory feedback will be provided during the tasks. The exercises will train both motor and cognitive functions.

SUMMARY:
The COVID-19 outbreak requires a rapid re-shaping of the entire organization of the rehabilitation services. This includes the design and planning of appropriate rehabilitation settings, intervention and logistics for organizing space for patients.

The aims of this study are: (a) to evaluate the feasibility of the bedside use of a novel rehabilitation device for upper limb in patients with stroke; (b) to evaluate the motor and cognitive outcomes of the treatment; (c) to validate the instrumental outcomes provided by the device.

DETAILED DESCRIPTION:
This study aims to:

1. evaluate the feasibility of the bedside use of a novel portable rehabilitation device for upper limb in patients with stroke in an inpatient setting;
2. assess motor and cognitive outcomes of the treatment;
3. validate the instrumental outcomes provided by the device.

Forty subacute stroke patients with upper limb hemiplegia will be enrolled. Patients' upper limb will be treated with a novel portable robotic device (Icone, Heaxel). The robot will be transferred to each patient's room, where the rehabilitation session will be performed, thanks to the portability of the device. During the treatment, patients will execute "exergames" involving elbow flexion-extension, shoulder protraction-retraction, internal-external rotation, flexion-extension and abduction-adduction. The exercises will be selected among the available ones to train both motor and cognitive functions. The rehabilitation intervention will include 30 rehabilitation sessions, each lasting 45 minutes, three to five times a week. In addition to the upper limb treatment, patients will receive a rehabilitation treatment for the lower limbs.

For Aim 1, the usability and the acceptability of the device and the satisfaction with the treatment will be evaluated at the end of the rehabilitation intervention by means of the System Usability Scale (SUS), the Technology Acceptance Model (TAM), and the Likert scale, respectively.

For Aim 2, the clinical effect of the treatment with the robot will be investigated by means of the following scales, assessed both at baseline and at discharge: the Fugl-Meyer Assessment for the upper extremity (FMA-UE), the Motricity Index (MI), the Modified Ashworth Scale (MAS), the Modified Barthel Index (mBI), the Numeric Pain Rating Scale (NPRS), and the Montreal Cognitive Assessment (MoCA)

For Aim 3, at baseline, each patient will perform the kinematic and kinetic assessment provided by the robot twice, one day apart, to assess the reliability of the kinematic parameters provided by the robot; moreover, the kinematic and kinetics assessment will be performed every ten rehabilitation sessions, to analyze the responsiveness of the kinematic parameters and possible "plateau" in the recovery process.

ELIGIBILITY:
Inclusion Criteria:

* first ischemic or hemorrhagic stroke (verified by MRI or CT);
* time latency within 6 months from stroke (subacute patients);
* age between 35-85 years;
* cognitive abilities adequate to understand the experiments and the follow instructions
* upper limb impairment (FMA-UE score ≤58);
* ability to give written consent;
* compliance with the study procedures.

Exclusion Criteria:

* history of recurrent stroke;
* inability to understand the instructions required for the study;
* fixed contractions in the affected limb (ankylosis, Modified Ashworth Scale equal to 4);
* severe deficits in visual acuity.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | After 30 rehabilitation sessions
  It is a tool for measuring the usability
Technology Acceptance Model (TAM) | After 30 rehabilitation sessions
  It is a tool for measuring the acceptability.
Likert Scale | After 30 rehabilitation sessions
  It is a tool for measuring the satisfaction.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment for upper extremity (FMA-UE) | At baseline; after 30 rehabilitation sessions
  The Fugl-Meyer Assessment is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment.
Motricity Index for the upper extremity (MI-UE) | At baseline; after 30 rehabilitation sessions
  It is a clinical instrument for characterizing the strength of the paretic upper extremity following stroke.
Modified Ashworth Scale (MAS) | At baseline; after 30 session rehabilitation sessions
  It is a clinical instrument for characterizing upper limb spasticity. Shoulder, elbow and wrist spasticity will be assessed.
Numeric Pain Rating Scale (NPRS) | At baseline; after 30 rehabilitation sessions
  It is a unidimensional measure of pain intensity in adults.
Modified Barthel Index (mBI) | At baseline; after 30 rehabilitation sessions
  It is a measure of independence in activities of daily living.
Montreal Cognitive Assessment (MoCA) | At baseline; after 30 rehabilitation sessions
  It is a widely used screening assessment for detecting cognitive impairment.
Kinematic parameters | At baseline (twice, one day apart); after 10 rehabilitation sessions; after 20 rehabilitation sessions; after 30 rehabilitation sessions
  The kinematics of the end-effector of the robot will be acquired during point-to-point tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Aprile, MD, PhD, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- Fondazione Don Carlo Gnocchi, Rome, Italy

IPD SHARING:
Plan to Share IPD: No